CLINICAL TRIAL: NCT03944317
Title: Randomized Controlled Trial of Azithromycin (AZ) and Sulphadoxine-pyrimethamine (SP) for Prophylaxis Against Malaria in Pregnancy (IPT)
Brief Title: Azithromycin (AZ) and Sulphadoxine-pyrimethamine (SP) for Malaria Prevention in Pregnant Women (IPT-AZ/IPT-SP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal Medical Centre, Owo (Industry)
Responsible Party: Principal Investigator, AHMED Ganiyu Olanipekun, Principal Investigator, Federal Medical Centre, Owo
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: FMCOWO
Record Dates: First submitted 2019-04-25; First posted 2019-05-09 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Malaria in Pregnancy; Pregnancy
Keywords: IPTip; SP; AZ
MeSH Terms: interventions — fanasil, pyrimethamine drug combination; Azithromycin

STUDY DESIGN:
Intervention Model Description: The design is a randomized comparative controlled study. Candidates for the study will be recruited from the antenatal booking clinic of our institution after being duly informed that participation is voluntary. Consented eligible pregnant woman will be recruited and those enrolled will be alloted into the two groups A and B of SP and Azithromycin respectively using a computer program (SPSS software version 21, Armonk, NY:IBM) generated sequence of numbers. Sequentially numbered sealed envelope containing either SP or AZ labelled will be allotted one after the other to participants. The personnel involved in the data collection and laboratory staff analyzing the samples will all not be aware of which group of patient is taking SP or Azithromycin while the doctors involved in administering the medication and the patients will be aware of which is being administered.
Who Masked: Outcomes Assessor
Masking Description: The personnel involved in the data collection and laboratory staff analyzing the samples will all not be aware of which group of patient is taking SP or Azithromycin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sulfadoxine pyrimethamine (Active Comparator): SP 1500/75mg tablet orally once starting from 16 weeks, at least at four weekly interval until delivery.
  Interventions: Drug: Sulfadoxine pyrimethamine
- Azithromycin (Active Comparator): A total of 1500mg Azithromycin tablets taken orally as 500mg daily for three consecutive days starting starting from 16weeks of pregnancy and to be repeated once at least after 4 weeks
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Sulfadoxine pyrimethamine — SP 1500/75mg tablet orally once starting from 16 weeks, at least at four weekly interval until delivery.
  Other Names: fansidar
  Arms: Sulfadoxine pyrimethamine
Drug: Azithromycin — A total of 1500mg Azithromycin tablets taken orally as 500mg daily for three consecutive days starting starting from 16weeks of pregnancy and to be repeated once at least after 4 weeks
  Other Names: Zithromax
  Arms: Azithromycin

SUMMARY:
AZITHROMYCIN VERSUS SULPHADOXINE-PYRIMETHAMINE FOR PROPHYLAXIS AGAINST MALARIA IN PREGNANCY IN OWO, SOUIHWESTERN NIGERIA: A RANDOMISED CONTROLLED TRIAL

OBJECTIVE: This study is to compare the efficacy of Azithromycin versus sulphadoxine-pyrimethamine as options of chemoprophylaxis against malaria in pregnancy.

METHOD: This is a randomized controlled trial with parallel assignment that will be conducted in the Obstetrics and Gynaecology department of the Federal Medical Centre. One hundred and sixty four (164) pregnant women who are eligible will be randomly allocated to 2 groups (A and B) of 84 each, using computer generated random numbers. Group A will receive sulfadoxine-pyrimethamine for malaria prophylaxis while Group B will receive azithromycin. All other aspects of antenatal care till delivery will be the same for all the women recruited. Maternal venous blood samples for malaria parasitaemia will be collected on recruitment and repeated at follow-up visits at any gestation there are symptoms of malaria; maternal peripheral blood film, placental and cord blood samples will be collected at delivery. All data will be documented in the data collection sheet. The results obtained will be subjected to statistical analysis using statistical package for social sciences (SPSS) version 21, Armonk, NY:IBM. The level of significance will be set at 5%. Outcomes will be compared across groups using Chi-square.

DETAILED DESCRIPTION:
Study design and Patient recruitment

The design is a randomized comparative controlled study. Candidates for the study will be recruited from the antenatal booking clinic of our institution after being duly informed that participation is voluntary. Informed consent will be obtained after the purpose, procedure, benefits, discomfort, risks and precautions associated with the study have been dully explained to them. Due diligence will be taken in adequately responding to any question or concern raised about the study. It will fully be explained to them that their participation is entirely voluntary. Also, if they are unwilling at any point to participate, they will be completely at liberty to discontinue their participation in the study which will not in any away affect their further and adequate management in the hospital. It will be explained that their participation in the study will not have any negative impact on them and their unborn babies and it has no financial benefits but the outcomes of the study may contribute to improved antenatal care. However, if there is additional financial cost (though not immediately foreseen) to any patient outside the cost of routine ANC visit, the investigator shall arrange for modest compensation. Consented eligible pregnant woman will be recruited and those enrolled will be alloted into the two groups A and B of SP and Azithromycin respectively using a computer program (SPSS software version 21, Armonk, NY:IBM) generated sequence of numbers. Sequentially numbered sealed envelope containing either SP or AZ labelled will be allotted one after the other to participants. The personnel involved in the data collection and laboratory staff analyzing the samples will all not be aware of which group of patient is taking SP or Azithromycin while the doctors involved in administering the medication and the patients will be aware of which is being administered.

ELIGIBILITY:
Inclusion Criteria:

* booked pregnant women
* Consent for the study
* Availability for follow-up during the pregnancy by keeping the next ANC appointment
* Willingness to deliver at the study site
* Age ≥ 18years
* comply with use of IPT-SP or Azithromycin medication as required by the study

Exclusion Criteria:

* Women treated for malaria in the index pregnancy
* Women who are severely ill (have medical conditions requiring hospital admission)
* Women who report prior adverse drug reaction to sulpha-containing medications and Azithromycin
* Patients with multiple gestations, sickle cell disease, HIV, IUGR and APH
* Women who did not want to participate in the study
* Age <18years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
malaria parasitaemia during pregnancy | through study completion, an average of 6 months
  number of pregnant women with maternal peripheral blood parasitaemia during pregnancy among pregnant women who use sulfadoxine pyrimethamine and azithromycin for malaria prevention in pregnancy

SECONDARY OUTCOMES:
malaria parasitaemia at the point of delivery | at the time of delivery
  number of pregnant women with maternal peripheral blood and placental parasitaemia, number of new born with cord blood parasitaemia at birth among pregnant women who use sulfadoxine pyrimethamine and azithromycin for malaria prevention in pregnancy

OTHER OUTCOMES:
low birth weight | at the time of delivery
  number of low birthweight babies among pregnant women who use sulfadoxine pyrimethamine and azithromycin for malaria prevention in pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Dr Aiyeyemi Adeyinka Joseph, MB;BS, FWACS, Study Director — Head of Department
Locations (1):
- FMCOWO, Owo, Ondo State, Nigeria

IPD SHARING:
Plan to Share IPD: No